CLINICAL TRIAL: NCT04890275
Title: Blood Flow Restricted Resistance Training in Peripheral Arterial Disease: a Randomised Controlled Trial Feasibility Study
Brief Title: Blood Flow Restricted Resistance Training in Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ER15905458
Record Dates: First submitted 2021-03-04; First posted 2021-05-18 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Blood flow restricted resistance exercise; Feasability
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR (Experimental): Participants will participate in a supervised low load lower body blood flow restriction resistance exercise program twice a week for 12 weeks
  Interventions: Other: Blood flow restricted resistance exercise (BFR)
- NON-BFR (Active Comparator): Participants will participate in a supervised low load lower resistance exercise program twice a week for 12 weeks (matched training volume as experimental arm but without BFR)
  Interventions: Other: Resistance exercise without blood flow restricted (NON-BFR)

INTERVENTIONS:
Other: Blood flow restricted resistance exercise (BFR) — Following a 5-minute low intensity warm-up, the BFR cuff will be placed at the most proximal portion of the leg inflated to 50% limb occlusion following standard BFR guidelines. Participants will then perform leg press including 1 set of 30 reps, then 3 sets of 15 reps at 20% 1RM. Rest for 5 minutes without cuff inflation. Cuffs will be re inflated and participants will perform knee extension including 3 x 15 repetitions at 20% 1RM.
  Arms: BFR
Other: Resistance exercise without blood flow restricted (NON-BFR) — Participants will follow the same exercise protocol as the blood flow restriction group but with out BFR.
  Arms: NON-BFR

SUMMARY:
A randomised controlled trial evaluating the feasibility and acceptability of a 12 week lower body blood flow restricted resistance exercise programme for people with peripheral arterial disease.

DETAILED DESCRIPTION:
The primary aim of this study is to determine the feasibility of 12 weeks of lower body resistance exercise performed with blood flow restriction (BFR) in people with peripheral arterial disease.

Resistance exercise with BFR involves placing inflatable cuffs proximal to the exercise limbs in order to manipulate blood flow and enhance the training response.

Secondary aim of this study is to evaluate changes in ABPI, muscle size, strength and physical function at mid-and post- intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with PAD 6 months post diagnosis.
* Ankle-brachial pressure index <0.9.
* People physically able to perform leg press and leg extension resistance exercise.

Exclusion Criteria:

* Ankle-brachial pressure index >0.89.
* People unable to visit the laboratory twice weekly for exercise sessions.
* People unable to do leg press and leg extension exercise.
* People whose walking is limited by a non-PAD condition.
* People with PAD with critical limb ischemia (including symptoms of pain at rest and skin ulcers).
* People with Dementia.
* People who have had major surgery or myocardial infarction within the past 6 months.
* Previous stroke.
* Previous thrombosis.
* People who have major surgery scheduled during the intervention period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Recruitment Rates | 3 months
  Defined as rate of invited participants who are eligible and consenting.
Retention Rates | 3 months
  Retention rates will be established as discontinuation with the exercise intervention and absence from the assessment sessions.
Acceptability of allocation | 3 months
  will be assessed by attrition rates, comparing participant withdrawal between experimental and control groups and reasons for dropout where appropriate.
Acceptability of the exercise study | 3 months
  Will be evaluated by participants feedback via one-to-one semi-structured interviews.
Completion Rates | 3 months
  Completion is determined by participants that attend baseline testing and post exercise intervention testing.

SECONDARY OUTCOMES:
Change in PAD severity | 3 months
  ankle-brachial pressure index
Change in muscle size | 3 months
  Size of vastus lateralis measured via ultrasound
Change in strength | 3 months
  Unilateral isometric maximal voluntary contraction
Change in walk ability | 3 months
  Measured via the 6-minute walk test
Change in physical function | 3 months
  Measured via timed up-and-go test

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Hallam University, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parkington T, Broom D, Maden-Wilkinson T, Nawaz S, Klonizakis M. Low-intensity resistance exercise with blood flow restriction for patients with claudication: A randomized controlled feasibility trial. Vasc Med. 2023 Dec;28(6):554-563. doi: 10.1177/1358863X231200250. Epub 2023 Oct 11. PMID 37819259